CLINICAL TRIAL: NCT07046897
Title: Analysis of the Gut Microbiota Composition After Consumption of Probiotic Bacteria
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Lund University, LTH
Record Dates: First submitted 2025-01-07; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Microbiota Analysis in Healthy Subjects
Keywords: Probiotics; Microbiota composition; Saliva; Faeces; Healthy individuals

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Consumption of probiotics strain 5 (Experimental): The participants will consume a probiotic product, a capsule with freeze-dries bacteria (B. coagulans strain 5).
  Interventions: Dietary Supplement: Consumption of probiotics strain 5
- Consumption of probiotics strain 6 (Experimental): The participants will consume a probiotic product, a capsule with freeze-dries bacteria (B. coagulans strain 6).
  Interventions: Dietary Supplement: Consumption of probiotics strain 6

INTERVENTIONS:
Dietary Supplement: Consumption of probiotics strain 5 — Consumption of probiotic capsules containing the probiotic bacteria Bacillus coagulans strain 5.
  Arms: Consumption of probiotics strain 5
Dietary Supplement: Consumption of probiotics strain 6 — Consumption of probiotic capsules containing the probiotic bacteria Bacillus coagulans strain 6.
  Arms: Consumption of probiotics strain 6

SUMMARY:
The goal of this intervention study is to evaluate the beneficial effect of the probiotic bacterium Bacillus coagulans in healthy volunteers. The main question it aims to answer is if the probiotic strains are modifying the microbiota composition in a beneficial way, evaluated in faecal- and saliva samples.

Primary hypothesis: The probiotic bacteria will modify the microbiota composition in faecal- and saliva samples.

Participants will consume the freeze-dried probiotic bacteria for 14 days. Before and after consumption, the participants will collect samples.

DETAILED DESCRIPTION:
Samples will be frozen immediately after collection and will be kept frozen until analysis at the Department of Process and Life Science Engineering, Faculty of Engineering, Lund University. For diversity measures, species identification and relative abundance of bacterial taxa, samples will be analysed by Illuminas MiSeq with the MiSeq reagent kit v3. Data will be analysed with bioinformatic pipeline QIIME2TM.

ELIGIBILITY:
Inclusion Criteria:

• You must be 18-65 years of age.

Exclusion Criteria:

* Participants must not be diagnosed with gastrointestinal diseases, autoimmune diseases or have diseases or medications that cause immune deficiency such as MS, type 1 diabetes, cancer or HIV.
* Participants must not have taken antibiotics in the month before or during the study.
* Participants must not consume other probiotic products or fermented foods during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
The gut microbiota composition | At enrollment and after 2 weeks of consumption.
  Diversity index will be calculated based on the results from next generation sequencing

SECONDARY OUTCOMES:
Relative abundance | At enrollment and after 2 weeks of consumption.
  Quantification of bacterial taxa will be calculated based on the results from next generation sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Åsa Håkansson, Associate Professor, Principal Investigator — Lund University, LTH
Locations (1):
- Department of Process and Life Science Engineering, Lund University, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No